CLINICAL TRIAL: NCT00586833
Title: The Role of Vascular Dysfunction in Limiting Cardiovascular Reserve in Patients With Heart Failure and a Preserved Ejection Fraction
Brief Title: Heart Failure and a Preserved Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Barry A. Borlaug, MD, Mayo Clinic
Other Study IDs: 07-001301; CHF
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Heart Failure
Keywords: Heart Failure; Heart Failure, Diastolic; Dyspnea, Paroxysmal; Edema, Cardiac
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic; Dyspnea, Paroxysmal; Edema, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood is drawn to evaluate BNP and cGMP pre and post exercise.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: No CHF/HTN Never diagnosed with CHF and undergoing current treatment for HTN
  Interventions: Procedure: O2 consumption max bike test
- 2: CHF with HFpEF HFpEF Cases will be recruited from the community. Subjects will be largely drawn from an existing Mayo database examining all incident cases of HF in Olmsted County.
  Interventions: Procedure: O2 consumption max bike test
- 3 Healthy normal adults: No identifiable cardiac issues at time of exercise.
  Interventions: Procedure: O2 consumption max bike test

INTERVENTIONS:
Procedure: O2 consumption max bike test — Single visit exercise study
  Other Names: Standard metabolic stress testing.; Pulmonary Capillary Blood Volume.; Plasma and Serum Neurohormone levels.; Ventricular data determined from echo-Doppler.; Vascular data obtained using a radial tonometry device

SUMMARY:
This will be a cross sectional study comparing patients with HFpEF and age-matched, non-HF controls recruited from the community. This design will allow for determination of biologically relevant differences in baseline ventricular and vascular function, and importantly, differences in the ability to augment ventricular and vascular function dynamically during exercise stress, when symptoms of HF typically are first noted. The endpoint of exercise-reserve function is novel and has been little examined in the existing HFpEF literature.

DETAILED DESCRIPTION:
Congestive heart failure (HF) is the leading cause of hospitalization among older Americans.1 Approximately half of affected patients have apparently normal systolic function (HF with preserved ejection fraction, HFpEF).2-4 In contrast to HF with low EF, there are no proven treatments for HFpEF, due largely to a lack of mechanistic understanding.4 HFpEF patients are typically older, hypertensive and female,2,3 and each of these characteristics is associated with vascular stiffening and dysfunction.5-7 Diastolic abnormalities may contribute to symptoms of exertional intolerance3,8, but non-cardiac limitations have recently been shown to be equally important.9-11 Patients with HFpEF display impaired decreases in mean vascular resistance in response to exercise, significantly limiting performance,9 yet this represents only one component of ventricular afterload. With aging and particularly in HFpEF, pulsatile load due to vascular stiffening and increased wave reflections becomes more magnified.6,12 The latter can be quantified by pulse wave velocity, arterial compliance and carotid augmentation index. These can be determined noninvasively, and while they have been shown to be abnormal in HFpEF patients at rest10,11, little is known about changes in each during exercise stress, or how this might modulate ventricular performance. Recent evidence indicates that endothelial and autonomic dysfunction are present in HFpEF9, but it is not known how these abnormalities might limit ventricular-vascular function with exercise. The primary objective of this proposal is to compare resting and exercise-induced changes in vascular function in patients with HFpEF and age-matched controls, to determine how these factors may affect exercise performance and cardiovascular reserve function.

Specific Aim 1. Contrast resting and exercise-induced changes in vascular stiffness, endothelial function, and afterload in patients with HFpEF to age-matched controls. Net, mean, and late components of afterload will be assessed by arterial elastance (Ea), systemic vascular resistance (SVR), and central augmentation index (AI). Vascular stiffness will be quantified by pulse wave velocity and total arterial compliance. Stiffness and afterload are dynamically modulated by endothelial and autonomic function, and these responses will be assessed by finger volume plethysmography. Parameters will be measured at rest, during upright cycle ergometry, and immediately post exercise by noninvasive blood pressure, tonometry and comprehensive echo-Doppler examination with tissue Doppler echo (TDE).

Specific Aim 2. Determine how baseline and exercise-induced changes in the vascular parameters measured in specific aim 1 are related to LV systolic and diastolic functional reserve, cardiac output response, metabolic exercise performance, and changes in pulmonary capillary blood volume. LV systolic and diastolic function will be assessed by echo-Doppler and TDE parameters at rest and immediately after peak exercise. Cardiac output response will be determined by the product of echo-Doppler stroke volume and heart rate. Exercise performance will quantified by expired gas analysis. Pulmonary blood volume will be estimated based upon the ratio of diffusion capacity of nitric oxide and carbon monoxide, obtained both at rest and immediately post exercise. Regression analyses will then be performed using the measured components of afterload and vascular stiffness as the independent variable and each of the above parameters as dependent output variables to delineate the role of vascular stiffening on exercise performance, reserve and ventricular-vascular coupling.

Specific Aim 3. Determine if vascular and ventricular stiffness properties measured in specific aim 1 are associated with abnormal neurohormonal responses to exercise. Blood samples will be obtained from HFpEF subjects and controls prior to and immediately after peak exercise to contrast exercise-induced changes in B-type natriuretic peptide levels and cyclic guanosine monophosphate levels.

ELIGIBILITY:
Inclusion Criteria:

* Consultation by a cardiologist for HF in the past 1 year
* (HF rigorously defined by the modified Framingham criteria9),
* able to exercise on a treadmill

Exclusion Criteria:

* decompensated HF; significant valvular disease; infiltrative, restrictive, or hypertrophic cardiomyopathy; cor pulmonale or significant pulmonary limitation; unstable coronary disease; atrial fibrillation; pregnancy; inability to exercise or suspend vasoactive medicines for at least 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HFpEF Cases will be recruited from the community. Subjects will be largely drawn from an existing Mayo database examining all incident cases of HF in Olmsted County.3 There are currently >350 pre-identified subjects with HFpEF from this study who may be eligible, which will greatly enrich the recruiting process.
  Control Subjects will be recruited from the community. Control subjects will be matched for age and gender to HFpEF subjects, but will have no history of HF hospitalization or significant exertional dyspnea suggestive of "preclinical" HF.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2007-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Contrast resting and exercise-induced changes in vascular stiffness, endothelial function, and afterload in patients with HFpEF to age-matched controls. | Throughout single visit.

SECONDARY OUTCOMES:
Determine how baseline and exercise-induced changes in the vascular parameters measured are related to LV systolic and diastolic functional reserve, cardiac output response, metabolic exercise performance, and changes in pulmonary cap | Throughout single visit
Determine if vascular and ventricular stiffness properties measured in specific aim 1 are associated with abnormal neurohormonal responses to exercise. | Immediately pre and post exercise

CONTACTS AND LOCATIONS:
Overall Officials: Barry A. Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States